CLINICAL TRIAL: NCT06047795
Title: Effect of Endurance Training On Functional Capacity and Quality of Life in Patients With Post-TB Lung Disease
Brief Title: Endurance Training in Patients With Post-TB Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rec/01657 Safa Marwa
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Tuberculosis; Post-Tuberculous Pleural Fibrosis; Post-Tuberculous Bronchiectasis
Keywords: Endurance training; Functional Capacity; Post-TB lung disease; Quality of Life
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Aerobic and respiratory endurance exercises with patient education
  Interventions: Other: Experimental
- Control (Placebo Comparator): Usual care (Patient Education, Home Plan)
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — Cycling 2 days per week with Borg dyspnea 4-6 level for 15-20 minutes/ day with 5 minutes warm-up and cool-down.
  Strengthening exercises for upper limb muscles (pull-ups and biceps curls) and for lower limb muscles (sit-to-stand and step-up exercises) with 3 sets of 8-12 repetitions * 2 days per week.
  Pursed Lip breathing exercise 3 sets of 5-10 repetitions for 6 weeks
  Arms: Interventional
Other: Control — Usual care: frontal chest radiographs, verbal advice to quit smoking, and reduce exposure to biomass smoke.
  Spirometry to screen for airway diseases. Antibiotic and systemic glucocorticoid therapy.
  Arms: Control

SUMMARY:
To determine the effects of endurance training on functional capacity and QOL(Quality of life) in patients with post-TB (tuberculosis) lung disease. Post-tuberculosis lung disease is a major health concern nowadays. There is limited evidence in the literature regarding the rehabilitation of patients with cured tuberculosis which leads to post-TB complications.

DETAILED DESCRIPTION:
Adults with post-TB respiratory symptoms experience skeletal muscle weakness due to inactivity, systemic inflammation, and poor nutrition, which is frequently made worse by poverty. Such patients experience a vicious cycle that includes decreased body weight, increasing morbidity, and higher mortality. People with Chronic Respiratory Diseases frequently avoid exercise, which causes them to lose motivation and decondition. This cycle of decline continues. In Pakistan, there is no concept of pulmonary rehabilitation for TB patients. The current study will attempt to fill this literature gap and also promote the concept of pulmonary rehabilitation for post-tuberculosis patients in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* TB (diagnosed) with Completed TB course
* Dyspnea (with or without cough)
* Age (18-50yrs).
* After 3 months of AFB and gene expert (-)
* Decreased PFT predicted values

Exclusion Criteria:

* Smoker, Diabetes, and cardiac patients
* Physical disabled, pregnant (lactating women)
* Sputum + testing for TB
* Gene expert
* CVD (unstable)
* Not willing to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Functional capacity | 3 weeks, 6 weeks
  Changes from baseline to 3 weeks and 6 weeks after the intervention, measured through 6 min walk test (6 MWT). It is a submaximal exercise test that can aid in assessing the functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters that an individual covers in 6 min without any support.
Dyspnea | 3 weeks, 6 weeks
  Changes from baseline to 3 weeks and 6 weeks after the intervention, measured through the BORG dyspnea scale. it uses a scale from 0 to 10, where 0 represents no dyspnea and 10 represents maximal dyspnea.
Forced Expiratory Volume in 1 second (FEV1) | 3 weeks,6 weeks
  Changes from the Baseline, the digital spirometer is used in the clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 3 weeks,6 weeks
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters
Peak Expiratory Flow (PEF) | 3 weeks,6 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Green Star NGO, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No